CLINICAL TRIAL: NCT06627166
Title: Clinical and Virological Characterization of Severe Acute Respiratory Infection Using PCR-Based Methods and Metagenomic Sequencing: a National Registry in Saudi Arabia
Brief Title: Viral Etiology of Severe Acute Respiratory InFection in CriticallY Ill Patients Registry
Acronym: VERIFY
Status: Terminated | Type: Observational
Why Stopped: Due to recruitment failure
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Dr Yaseen Arabi, Chairman intensive care unit, King Abdullah International Medical Research Center
Other Study IDs: RC20-294-R
Record Dates: First submitted 2023-03-12; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-04

CONDITIONS: Severe Acute Respiratory Infection
Keywords: SARI; Critically ill; Infection; viruses
MeSH Terms: conditions — Critical Illness; Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swab, MINI BAL samples, Serum samples, Plasma sample, and Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe Acute Respiratory Infection (SARI): Nasopharyngeal swab, MINI BAL samples, Serum samples, Plasma sample, and Blood sample (RNA) will be collected from patients on day 0 (baseline) of enrollment, and on day 14 of enrollment.
  SAMPLING PROCEDURES:
  1. Nucleic acid extraction
  2. Polymerase chain reaction (PCR) 2.1 Testing for MERS-CoV will be performed by RT-PCR 2.2 We will test for Infleunza H and N PCR for influenza H 2.3 We will also test for a panel of viruses using PCR multiplex that includes influenza A ; influenza B ; influenza C ; influenza A (H1N1) swl ; parainfluenza viruses 1, 2, 3 and 4 ; coronaviruses NL63, 229E, OC43 and HKU1; human metapneumoviruses A/B; rhinovirus ;respiratory syncytial viruses A and B; adenovirus; enterovirus; parechovirus; bocavirus.
  3.16S PCR and sanger sequencing for bacterial detection 4.Metagenomics /Next Generation Sequencing 5.Microbiome bioinformatics analysis

SUMMARY:
SARI is a major public health problem in Saudi Arabia and leads to considerable morbidity and mortality. Most SARI-related mortality occurs in patients admitted to ICUs across the country. RVIs alone and as precipitating causes of bacterial co-infections are under-recognized as causes of critical SARI. Therefore, data regarding the role of RVIs in critically ill patients with SARI in Saudi Arabia are greatly needed to fill the current gaps with respect to pathogens, disease pathogenesis, current treatment approaches, and clinical outcomes.

In the VERIFY multicenter national registry, we aim to determine the viral etiologies of SARI in mechanically ventilated critically ill patients. We aim to collect inventory samples (blood, and nasopharyngeal swabs, mini BAL) from >10 sites in Saudi Arabia from different regions to enhance generalizability of data.

DETAILED DESCRIPTION:
Data on the burden, severity and etiology of SARI amongst critically ill patients will be expected to be of a great value in guiding the prioritization of prevention and control efforts18 and in the design of future intervention studies of antivirals and other therapeutic modalities.

Because influenza is a common cause of serious respiratory illness in Saudi Arabia, although only limited data are available on the most severely ill patients with influenza, we will conduct surveillance in SARI critically ill patients and perform typing and subtyping of influenza viruses in BAL samples. We will store samples for future examination of predisposing risk factors including genetic factors.

Multiplex PCR will reduce the cost and time to detect the respiratory pathogens. In recent years, the falling costs of Whole Genome Sequencing (WGS) technologies have has proven to be a valuable tool to understand the growing threat of emerging pathogens. Metagenomic next-generation sequencing (M-NGS) has transformative effect in the last decade to investigate and understand complex microbial communities. M-NGS is simply capturing and determining all nucleic acids in a sample which allowed to identify a mixed population of microorganisms. This powerful platform simultaneously identifies genetics materials of any organisms unbiased to other methods that used specific primers to identify specific targets.

The primary objective of the VERIFY registry is to examine the virological etiologies of SARI among mechanically ventilated critically ill patients in a geographical representative sample from Saudi Arabia in order to obtain a better estimate of viral pathogen prevalence by systematic lower respiratory tract sampling and use of serology among critically ill patients in a geographical representative sample from Saudi Arabia. Contribution of viruses may be under-estimated due to the use of upper respiratory tract specimens only, and late presentation of cases to ICU (at which time antigen is no longer detectable). Therefore a systematic approach using mini-BAL to obtain lower respiratory samples will likely yield better estimate.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥14 years old) patients
* A clinical presentation consistent with community-acquired SARI/pneumonia
* AND admitted to the ICU because of respiratory failure or sepsis
* AND is invasively mechanically ventilated.

Exclusion Criteria:

* Diagnosed with COVID-19
* Duration of illness > 14 days since symptom onset
* Did not meet inclusion criteria in the first 48 hrs of admission to the ICU.
* Patient already enrolled in the study
* Participant or legal guardian refuses to participate in the study.
* Diagnosis is not related to SARI
* Enrolled in interventional trial of investigational therapeutics for pneumonia.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients with SARI in critical care setting.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of different viral and bacterial pathogens among critically ill patients with SARI | 14 Days
  Viral pathogens include influenza virus and MERS corona virus

SECONDARY OUTCOMES:
Clinical features and response to treatment of SARI of different etiologies. | 90 days
  Clinical data collection include demographic (Age in years, BMI in kg/m^2)
Clinical features and response to treatment of SARI of different etiologies. | 90 days
  Risk factors (Admission diagnosis, smoking, chronic comorbidities)
Clinical features and response to treatment of SARI of different etiologies. | 90 days
  Clinical course in the ICU (mechanical ventilation, vasopressor use, renal replacement therapy, tracheostomy)
Clinical features and response to treatment of SARI of different etiologies. | 90 days
  outcomes (90 day mortality, ICU length of stay, hospital length of stay, mechanical ventilation duration)

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen Arabi, Principal Investigator — King Abdulaziz Medical City
Locations (1):
- Intensive Care Department, King Abdulaziz Medical City, National Guard Health Affairs, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huai Y, Guan X, Liu S, Uyeki TM, Jiang H, Klena J, Huang J, Chen M, Peng Y, Yang H, Luo J, Zheng J, Peng Z, Huo X, Xiao L, Chen H, Zhang Y, Xing X, Feng L, Hu DJ, Yu H, Zhan F, Varma JK. Clinical characteristics and factors associated with severe acute respiratory infection and influenza among children in Jingzhou, China. Influenza Other Respir Viruses. 2017 Mar;11(2):148-156. doi: 10.1111/irv.12419. Epub 2016 Sep 20. PMID 27465959
- [Background] Nguyen HKL, Nguyen SV, Nguyen AP, Hoang PMV, Le TT, Nguyen TC, Hoang HT, Vuong CD, Tran LTT, Le MQ. Surveillance of Severe Acute Respiratory Infection (SARI) for Hospitalized Patients in Northern Vietnam, 2011-2014. Jpn J Infect Dis. 2017 Sep 25;70(5):522-527. doi: 10.7883/yoken.JJID.2016.463. Epub 2017 Mar 28. PMID 28367882
- [Background] Meerhoff TJ, Simaku A, Ulqinaku D, Torosyan L, Gribkova N, Shimanovich V, Chakhunashvili G, Karseladze I, Yesmagambetova A, Kuatbayeva A, Nurmatov Z, Otorbaeva D, Lupulescu E, Popovici O, Smorodintseva E, Sominina A, Holubka O, Onyshchenko O, Brown CS, Gross D. Surveillance for severe acute respiratory infections (SARI) in hospitals in the WHO European region - an exploratory analysis of risk factors for a severe outcome in influenza-positive SARI cases. BMC Infect Dis. 2015 Jan 8;15:1. doi: 10.1186/s12879-014-0722-x. PMID 25567701
- [Background] Ruuskanen O, Lahti E, Jennings LC, Murdoch DR. Viral pneumonia. Lancet. 2011 Apr 9;377(9773):1264-75. doi: 10.1016/S0140-6736(10)61459-6. Epub 2011 Mar 22. PMID 21435708